CLINICAL TRIAL: NCT01170377
Title: The Effect of Valproate on the Required Dose of Propofol for Sedation in Patients With Mental Retardation
Brief Title: Effect of Valproate on Propofol
Status: Completed | Type: Observational
Sponsor: Okayama University (Other)
Responsible Party: Department of Dental Anesthesiology and Special Care Dentistry, Okayama University Graduate School of Medicine, Dentistry and Pharmaceutical Sciences
Other Study IDs: 141mina
Record Dates: First submitted 2010-07-21; First posted 2010-07-27 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2010-08

CONDITIONS: Mental Retardation
Keywords: Intravenous sedation; Dental treatment; Mental retardation; Antiepileptic drug; Valproate; Propofol
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mental Retardation: Patients receiving valproate or not

SUMMARY:
The aim of this study is to evaluate the effect of valproate on the required dose of propofol for sedation in patients with mental retardation.

DETAILED DESCRIPTION:
The intravenous sedation with propofol is very useful for patients with mental retardation and challenging behavior. However, it is very difficult to titrate the dose of propofol for maintaining the adequate sedation depth because of the difficulty of verbal communication with them. Most of them have a epilepsy and take antiepileptic drugs. Antiepileptic drugs are thought to influence on the effect of anesthetics. Valproate is reported to inhibit the metabolism of propofol. Therefore, we divide the patients into two groups : patients receiving valproate (valproate group), patients receiving no antiepileptic drugs (control group), and compare the required dose of propofol and the recovery time.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 16 or over
2. American Society of Anesthesiologists (ASA) physical status 1 or 2
3. The treatment of dental caries, endodontics, periodontics and prosthesis were planed
4. Participants had moderate or severe Mental Retardation, and were not completely cooperated with dental treatment

Exclusion Criteria:

1. Patients could communicate and cooperate with dental treatment, but used dental sedation for decrease of the anxiety and the fear about dental treatment or another reasons
2. Patients needed premedication and inhalational anesthetics
3. Patients had uncontrolled or sever medical condition

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with mental reterdation
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The dose of anesthesia agent | 1 day
The recovery time of eyelash reflex | 1 day
The recovery time of eye opening | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Minako Ishii, D.D.S., Principal Investigator — Department of Dental Anesthesiology and Special Care Dentistry, Okayama University Graduate School of Medicine, Dentistry and Pharmaceutical Sciences
Locations (1):
- Department of Dental Anesthesiology and Special Care Dentistry, Okayama University Graduate School of Medicine, Dentistry and Pharmaceutical Sciences, Okayama, Japan